CLINICAL TRIAL: NCT03040102
Title: Randomized Study of a Hospice Video Educational Tool for Patients With Advanced Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Areej El-Jawahri, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-026
Record Dates: First submitted 2017-01-28; First posted 2017-02-02 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospice Video Educational Tool (Experimental): * The hospice video educational tool is a 6 minute video
  * Participants will watch an approximately 6-minute digital video regarding hospice on an iPad
  Interventions: Other: Hospice Video Educational Tool
- Hospice Verbal Narrative (Active Comparator): * The RA will read a verbal narrative that is identical to the narrative of the video to participants
  * Standard of Care practice is used
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Hospice Video Educational Tool — it's a 6 minute video regarding hospice care
  Arms: Hospice Video Educational Tool
Other: Standard of Care — Standard of Care practice is used
  Arms: Hospice Verbal Narrative

SUMMARY:
The purpose of this research study is to compare two ways to educate patients with cancer and their caregivers about hospice care services

DETAILED DESCRIPTION:
The purpose of this research study is to compare two ways to educate patients with cancer and their caregivers about hospice care services - a video educational tool or a verbal narrative. The study will assess the effect of these methods on patients' and caregivers' knowledge about hospice care, as well as their perceptions and preferences for this service.

Using this research, the investigators hope to find out the best way to help patients and their loved ones better understand hospice care. The educational methods used in this study (the video educational tool or verbal narrative) are meant to serve as an introduction to hospice care. Further details about hospice should be discussed directly with your care team.

This study will enroll 150 patients with advanced cancer and up to 150 of their caregivers in this randomized clinical trial. The study will use questionnaires to measure the participant and the caregivers' knowledge of hospice care, as well as your perceptions and preferences for these services. Study assessments will be completed before and after watching the video or hearing the verbal narrative in the hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients Eligibility Criteria:

* Adult patients (≥18 years) with a diagnosis of metastatic solid cancer.
* A prognosis of 12 months or less based on the treating oncologist's assessment.
* The ability to provide informed consent.
* Ability to comprehend and speak English.

Caregivers Eligibility Criteria:

* Adult caregivers (>18 years) of patients who have agreed to participate in study.
* A relative or a friend upon whom the patient relies for help and who will be likely to be present during hospitalization, or willing to participate by phone.
* Ability to comprehend and speak English.

Exclusion Criteria:

Patients Exclusion Criteria:

-Significant uncontrolled psychiatric disorder (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the treating clinician believes prohibits the ability to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Patient Preference for Hospice Question | immediately after the video intervention or verbal narrative
  We will ask patients whether they would prefer to receive hospice care at the end of life (yes vs. no)

SECONDARY OUTCOMES:
Patient knowledge about hospice Questionnaire | immediately after the video intervention or verbal narrative
  we will assess knowledge about hospice using 10 knowledge questions

OTHER OUTCOMES:
Patient Perception of Hospice Care Questionnaire | immediately after the video intervention or verbal narrative
  we will assess perception of hospice using the Hospice Perception Questionnaire
Patient Hospice Utilization | 1 year after study completion
  We will assess patient hospice utilization and length of stay in hospice
Caregiver Preference for Hospice Question | immediately after the video intervention or verbal narrative
  we will assess caregiver's preference for their loved one using hospice (yes vs. no)
Caregiver Knowledge about Hospice Questionnaire | immediately after the video intervention or verbal narrative
  we will assess knowledge about hospice using 10 knowledge questions
Caregiver Perception of Hospice Care Questionnaire | immediately after the video intervention or verbal narrative
  we will assess perception of hospice using the Hospice Perception Questionnaire
Caregiver satisfaction with end-of-life care (FAMCARE) | 1 year after study completion
  We will use 9 items from the FAMCARE to assess caregivers' satisfaction with patient's end of life care

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No